CLINICAL TRIAL: NCT07074145
Title: WEAVE NM Project: Heart Health and Nutrition for Life (HHNL)
Brief Title: WEAVE NM: Heart Health and Nutrition for Life
Acronym: WEAVE HHNL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Westat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sub-OTA 6922-03-COVID-S014; OT2HL158287 (NIH)
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: Hypertension; Community Health Worker; Health Education; Blood Pressure
MeSH Terms: conditions — Hypertension; Health Education | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Drawing on methodological innovations in the design of community-partnered research and randomized controlled trials, this study will use a multi-wave, two-arm randomized controlled trial with two study phases and an active control condition to measure the effectiveness of the HHNL expanded primary care intervention as compared to First Nations Community HealthSource (FNCH) standard clinical care for hypertension, alongside supported blood pressure self-monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HHNL Educational Interventional Arm (Experimental): Arm 1 of this study will consist of individuals initially assigned to the HHNL educational intervention, alongside FNCH standard care with blood pressure self-monitoring, to assess improvements in systolic blood pressure outcomes relative to those initially assigned to FNCH standard care with blood pressure self-monitoring only (Arm 2). The educational intervention is received in the first 6 months for participants within Arm 1.
  Interventions: Behavioral: Heart Health and Nutrition for Life (HHNL); Behavioral: Self-Measured Blood Pressure
- Comparator Arm: Standard of Care and Self Blood Pressure Monitoring (Active Comparator): Arm 2 will serve as the active control condition of FNCH standard care supplemented with supported self-measured blood pressure (SMBP). SMBP, itself, is an evidence-based intervention. Inclusion of an active control in this study is designed to facilitate both enhanced participant benefit and enhanced science, while allowing the investigators to assess the add-on impacts of the HHNL expanded primary care intervention more rigorously. Arm 2 receives the educational intervention within the second 6 months of study participation.
  Interventions: Behavioral: Self-Measured Blood Pressure

INTERVENTIONS:
Behavioral: Heart Health and Nutrition for Life (HHNL) — The CHW-led educational intervention will draw on two evidence-based programs, Healthy for Life (American Heart Association) and Your Heart, Your Life (NHLBI). Both curricula are designed to be facilitated by community health workers/promotores de salud and have been tested in both English and Spanish. Study-adapted curricular elements will include 12 core educational activities, delivered in six, two-hour, in-person sessions. In the context of expected family and work obligations alongside limited resources of FNCH patients, the investigators anticipate structuring sessions over, at most, 2 months with a class size of approximately 5-15 patients. In the CHW-led educational intervention, participants will learn about topics such as understanding risk for heart disease, the importance of physical activity, affordable healthy eating, and how family members can support health.
  Arms: HHNL Educational Interventional Arm
Behavioral: Self-Measured Blood Pressure — Self-measured blood pressure (SMBP) is a proven, cost-effective strategy to improve blood pressure control by promoting patient engagement and medication adherence. All study participants will receive the same validated BP monitor, with cuff sizes adjusted as needed, selected from the US Blood Pressure Validated Device Listing. Patients will be trained using the AMA's 7-Step SMBP Quick Guide, consistent with FNCH clinical education practices. They will be asked to record baseline BP readings and complete at least one SMBP cycle per month during the 12-month study. Each cycle includes at least three consecutive days of morning and evening BP measurements.

SUMMARY:
WEAVE NM (Wide Engagement for Assessing Vaccine Equity in New Mexico) is a community-based research initiative working to improve health outcomes in underserved populations, with a current focus on hypertension and food justice. The project centers on the lived experiences of Native American, African American, Hispanic/Latino, and Asian American residents in Albuquerque's International District and South Valley. With guidance from community voices and ongoing collaboration with local organizations, health providers, and residents, the initiative integrates cultural values, public policy, and social realities into solutions that promote equity and wellness.

As part of this work, a clinical trial is being conducted through First Nations Community HealthSource (FNCH) to evaluate a culturally tailored blood pressure intervention called Heart Health and Nutrition for Life (HHNL). The trial includes patients who receive standard hypertension care and blood pressure self-monitoring, with one group also participating in a community health worker-led educational program in their first six months of study enrollment. This curriculum addresses healthy eating, physical activity, medication adherence, stress reduction, and avoidance of alcohol and tobacco, all delivered with cultural sensitivity and community insight. After six months, the groups switch roles, allowing all participants to receive the education component.

Participants' progress is measured over a 12-month period by tracking changes in blood pressure, cholesterol, weight, blood sugar (HbA1c), and emotional well-being. The aim is to determine whether this community-supported approach improves outcomes more effectively than standard care alone with blood pressure self-monitoring. This study represents a broader effort to create long-term, community-rooted solutions to chronic health issues by addressing the social and environmental factors that influence well-being.

For individuals living in the International District or South Valley, this project offers the opportunity to take part in research that respects cultural identity and prioritizes real-world impact on health. Interested patients and families can contact their provider at FNCH to learn more about participation.

DETAILED DESCRIPTION:
HHNL is a two-arm, randomized, controlled trial with two study phases and an active control condition, enrolling 240 adults with hypertension from First Nations Community HealthSource (FNCH), including Native American, Latinx, African American, and Asian American participants. All receive education, blood pressure monitors, and study questionnaires.

This clinical trial component is designed to evaluate whether a healthy lifestyle program led by community health workers-called Heart Health and Nutrition for Life (HHNL)-improves blood pressure control more effectively than standard care with blood pressure self-monitoring alone. The HHNL program includes blood pressure self-monitoring and culturally tailored education sessions. The trial is being conducted with patients receiving care at First Nations Community HealthSource (FNCH), a federally qualified health center serving a varying population in Albuquerque, New Mexico.

Participants are randomly assigned to one of two groups. One group receives the HHNL education program in their first six months of study enrollment, along with FNCH's standard care and blood pressure self-monitoring. The other group receives standard care and blood pressure self-monitoring alone for the first six months, after which they receive the HHNL education program in their second six months of study enrollment. The goal is to compare outcomes over time and between groups to understand the added value of the HHNL program.

The primary focus is on changes in systolic blood pressure over the first six months. Data will be collected at baseline, 3-4 months, and six months to track progress, with data at 3-4 months allowing early insights following the conclusion of the education sessions.

In addition to systolic blood pressure, the study will also examine other health indicators, including diastolic blood pressure, lipid levels (total cholesterol, LDL, HDL, and triglycerides), HbA1c, body mass index (BMI), and psychological distress. Researchers will also assess behavior-related factors such as medication adherence, blood pressure monitoring habits, physical activity, healthy eating, alcohol and tobacco use, and perceptions of health risks and benefits. These outcomes will be analyzed from baseline to six months, with a focus on comparing the two groups and understanding the immediate effects of the intervention.

Over the full 12-month study period, the research team expects to see specific trends within each group. For those starting with the HHNL education program, improvements in health outcomes are anticipated in the first six months, with those gains maintained after transitioning to standard care with blood pressure self-monitoring alone. For participants who begin with standard care with blood pressure self-monitoring alone and later receive the HHNL educational sessions, improvements are expected primarily during the second half of the study.

The trial is being developed and implemented with ongoing input from a Community Advisory Council to ensure cultural relevance, community alignment, and consistent guidance of the research process.

ELIGIBILITY:
Inclusion Criteria:

* Currently a FNCH patient or are willing and able to become a FNCH patient
* Current diagnosis of hypertension that was not onset due to pregnancy
* Able to speak and read English or Spanish
* Cognitively and physically able to independently understand and complete study procedures and provide written informed consent
* Self-report at least one systolic blood pressure reading of 130 or greater in the last six months OR show a systolic blood pressure reading of 130 or greater in baseline screening
* Live in and receive mail in Albuquerque, New Mexico

Exclusion Criteria:

* By design, adults unable to consent, individuals not yet adults, and prisoners will not be included in this study.
* Patients who self-report pregnancy will be automatically excluded from the study. While the investigators are not systematically screening for pregnancy throughout the study, if an individual self-reports pregnancy during the study, they will be withdrawn from study participation and offered the opportunity to re-join the study once no longer pregnant, if activities are still available, following general study procedures.
* Individuals who are not able to complete study procedures due to mental or behavioral health conditions, incarceration, or inability to physically bear an arm cuff will also be excluded from the study.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Baseline measurement and at about 3-, 6-, and 12- month timepoints
  Clinically measured blood pressure levels

SECONDARY OUTCOMES:
Diastolic Blood Pressure | Measured at baseline and at about 3-, 6-, and 12-month timepoints.
  Clinically measured diastolic blood pressure
HbA1c | Months 0, 3, 6 & 12
  Diabetes Indicator
BMI | Months 0, 3, 6 & 12
  Body Mass Index
Lipid levels (total cholesterol, LDL, HDL, triglycerides) | Months 0, 3, 6 & 12
  Cholesterol
Psychological Distress | Months 0, 3, 6 & 12
  Kessler Psych Distress scale (K10)

OTHER OUTCOMES:
Consistency of BP self-monitoring | Monthly: Months 1-12
  Monthly self-measured BP logs
Adherence to anti-HTN medication | Months 0, 3, 6 & 12
  H-SCALE subscale
Healthy eating | Months 0, 3, 6 & 12
  H-SCALE subscale
Physical Activity Engagement | Months 0, 3, 6 & 12
  H-SCALE subscale
Weight management | Months 0, 3, 6 & 12
  H-SCALE subscale
Avoiding alcohol and tobacco | Months 0, 3, 6 & 12
  H-SCALE subscale
Self-efficacy | Months 0, 3, 6 & 12
  Health Belief Model adapted subscale
Perceived susceptibility | Months 0, 3, 6 & 12
  Health Belief Model adapted subscale
Perceived severity | Months 0, 3, 6 & 12
  Health Belief Model adapted subscale
Perceived benefits | Months 0, 3, 6 & 12
  Health Belief Model adapted subscale
Community pride | Months 0, 3, 6 & 12
  Adapted single-item behavior change influence outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tassy Parker, PhD, RN, Principal Investigator — University of New Mexico; Linda Son-Stone, Ed D, MPH, Principal Investigator — First Nations Community HealthSource; Lisa Cacari Stone, PhD, MS, MA, Principal Investigator — University of New Mexico
Locations (1):
- First Nations Community HealthSource, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified repository will house all data shared with Westat, minus identifiers (e.g., birth month, detailed geographic data), and include additional variables such as BP, BMI, psychological distress, medication adherence, lifestyle behaviors, perceptions, community pride, family cohesion, spiritual practices, and healthcare discrimination.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Scientific data generated during WEAVE NM HHNL will be deposited by the end of the proposed grant funding period or by time of associated publication, whichever comes first. Archiving practices of the chosen data repository will support standardized back up and replication, and all shared scientific data will remain deposited with ongoing monitoring for accessibility for a minimum of three years after the end of the grant funding period.
Access Criteria: The WEAVE NM HHNL project is expected to generate individual-level clinical data and self-reported health and process data. This data will be preserved and shared at the unit-of-observation level when permitted by federal, state, local, or Tribal law and where participant privacy and community safety can be maintained. All quantitative data will be de-identified using best practices outlined in the Inter-university Consortium for Political and Social Research's (ICPSR) Guide to Social Science Data Preparation and Archiving, 6th edition, and by applying the HIPAA Safe Harbor method to remove all 18 identifiers from datasets containing protected health information. Accompanying metadata will ensure the data can support both validation of findings and the generation of new analyses. Supporting documentation will include key metadata elements such as study protocols, data collection instruments, and study description.

REFERENCES:
- [Background] Kandzari DE, Mahfoud F, Weber MA, Townsend R, Parati G, Fisher NDL, Lobo MD, Bloch M, Bohm M, Sharp ASP, Schmieder RE, Azizi M, Schlaich MP, Papademetriou V, Kirtane AJ, Daemen J, Pathak A, Ukena C, Lurz P, Grassi G, Myers M, Finn AV, Morice MC, Mehran R, Juni P, Stone GW, Krucoff MW, Whelton PK, Tsioufis K, Cutlip DE, Spitzer E. Clinical Trial Design Principles and Outcomes Definitions for Device-Based Therapies for Hypertension: A Consensus Document From the Hypertension Academic Research Consortium. Circulation. 2022 Mar 15;145(11):847-863. doi: 10.1161/CIRCULATIONAHA.121.057687. Epub 2022 Mar 14. PMID 35286164
- [Background] Ma C. An investigation of factors influencing self-care behaviors in young and middle-aged adults with hypertension based on a health belief model. Heart Lung. 2018 Mar-Apr;47(2):136-141. doi: 10.1016/j.hrtlng.2017.12.001. Epub 2018 Feb 1. PMID 29395265
- [Background] Khorsandi M, Fekrizadeh Z, Roozbahani N. Investigation of the effect of education based on the health belief model on the adoption of hypertension-controlling behaviors in the elderly. Clin Interv Aging. 2017 Jan 27;12:233-240. doi: 10.2147/CIA.S117142. eCollection 2017. PMID 28184154
- [Background] Warren-Findlow J, Krinner LM, Vinoski Thomas E, Coffman MJ, Gordon B, Howden R. Relative and Cumulative Effects of Hypertension Self-Care Behaviors on Blood Pressure. West J Nurs Res. 2020 Mar;42(3):157-164. doi: 10.1177/0193945919851111. Epub 2019 May 26. PMID 31130078
- [Background] Carey RM, Whelton PK; 2017 ACC/AHA Hypertension Guideline Writing Committee. Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Synopsis of the 2017 American College of Cardiology/American Heart Association Hypertension Guideline. Ann Intern Med. 2018 Mar 6;168(5):351-358. doi: 10.7326/M17-3203. Epub 2018 Jan 23. PMID 29357392
- [Background] Rink E, Knight K, Ellis C, McCormick A, FireMoon P, Held S, Webber E, Adams A. Using Community-Based Participatory Research to Design, Conduct, and Evaluate Randomized Controlled Trials with American Indian Communities. Prev Chronic Dis. 2020 Nov 12;17:E143. doi: 10.5888/pcd17.200099. PMID 33180688
- [Background] Kwon SC, Tandon SD, Islam N, Riley L, Trinh-Shevrin C. Applying a community-based participatory research framework to patient and family engagement in the development of patient-centered outcomes research and practice. Transl Behav Med. 2018 Sep 8;8(5):683-691. doi: 10.1093/tbm/ibx026. PMID 30202926
- [Background] U.S. Department of Health and Human Services. (2008). Your heart, your life: A community health worker's manual. NHLBI. https://www.nhlbi.nih.gov/files/docs/resources/heart/lat_mnl_en.pdf
- [Background] Healthy for Life. www.heart.org. (n.d.). https://www.heart.org/en/healthy-living/companycollaboration/healthy-for-life.
- [Background] Moore KR, Schroeder EB, Goodrich GK, Manson SM, Malone AS, Pieper LE, Son-Stone L, Johnson D, Steiner JF. Racial and Ethnic Equity in Care for Hypertension and Diabetes in an Urban Indian Health Organization. J Racial Ethn Health Disparities. 2023 Jun;10(3):1319-1328. doi: 10.1007/s40615-022-01317-3. Epub 2022 May 3. PMID 35503165
- [Background] Schroeder EB, Moore K, Manson SM, Baldwin MA, Goodrich GK, Malone AS, Pieper LE, Xu S, Fort MM, Johnson D, Son-Stone L, Steiner JF. An Interactive Voice Response and Text Message Intervention to Improve Blood Pressure Control Among Individuals With Hypertension Receiving Care at an Urban Indian Health Organization: Protocol and Baseline Characteristics of a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2019 Apr 2;8(4):e11794. doi: 10.2196/11794. PMID 30938688
- [Background] Meador M, Hannan J, Roy D, Whelihan K, Sasu N, Hodge H, Lewis JH. Accelerating Use of Self-measured Blood Pressure Monitoring (SMBP) Through Clinical-Community Care Models. J Community Health. 2021 Feb;46(1):127-138. doi: 10.1007/s10900-020-00858-0. PMID 32564288
- [Background] Stupplebeen DA, Pirkle CM, Sentell TL, Nett BMI, Ilagan LSK, Juan B, Medeiros J, Keliikoa LB. Self-Measured Blood Pressure Monitoring: Program Planning, Implementation, and Lessons Learned From 5 Federally Qualified Health Centers in Hawai'i. Prev Chronic Dis. 2020 Jun 25;17:E47. doi: 10.5888/pcd17.190348. PMID 32584755
- [Background] Blue Bird Jernigan V, D'Amico EJ, Duran B, Buchwald D. Multilevel and Community-Level Interventions with Native Americans: Challenges and Opportunities. Prev Sci. 2020 Jan;21(Suppl 1):65-73. doi: 10.1007/s11121-018-0916-3. PMID 29860640
- [Background] Parker T, Kelley A, Cooeyate N, Tsosie N. Tribal Perspectives on Hypertension: Results From the Center for Native American Health Native-CHART Needs Assessment. J Prim Care Community Health. 2022 Jan-Dec;13:21501319221144269. doi: 10.1177/21501319221144269. PMID 36524696
- [Background] Sanchez V, Cacari Stone L, Moffett ML, Nguyen P, Muhammad M, Bruna S, Urias-Chauvin R. Process evaluation of a promotora de salud intervention for improving hypertension outcomes for Latinos living in a rural U.S.-Mexico border region. Health Promot Pract. 2014 May;15(3):356-64. doi: 10.1177/1524839913516343. Epub 2014 Jan 6. PMID 24396118
- [Background] Cacari Stone L, Sanchez V, Bruna SP, Muhammad M, Zamora Mph C. Social Ecology of Hypertension Management Among Latinos Living in the U.S.-Mexico Border Region. Health Promot Pract. 2022 Jul;23(4):650-661. doi: 10.1177/1524839921993044. Epub 2021 Mar 12. PMID 33709805
- [Background] Baker EA, Barnidge EK, Schootman M, Sawicki M, Motton-Kershaw FL. Adaptation of a Modified DASH Diet to a Rural African American Community Setting. Am J Prev Med. 2016 Dec;51(6):967-974. doi: 10.1016/j.amepre.2016.07.014. Epub 2016 Sep 12. PMID 27633485
- [Background] Steinberg D, Kay M, Burroughs J, Svetkey LP, Bennett GG. The Effect of a Digital Behavioral Weight Loss Intervention on Adherence to the Dietary Approaches to Stop Hypertension (DASH) Dietary Pattern in Medically Vulnerable Primary Care Patients: Results from a Randomized Controlled Trial. J Acad Nutr Diet. 2019 Apr;119(4):574-584. doi: 10.1016/j.jand.2018.12.011. PMID 30905430